CLINICAL TRIAL: NCT03973541
Title: EXPOSURE IN VIRTUAL REALITY FOR SOCIAL ANXIETY DISORDER - A Randomized Controlled Superiority Trial Comparing Cognitive Behavioral Therapy With Virtual Reality Based Exposure to Cognitive Behavioral Therapy With in Vivo Exposure.
Brief Title: CBT With VR Based Exposure for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Collaborators: Universite du Quebec en Outaouais (Other)
Responsible Party: Principal Investigator, Per T Ørskov, PhD, Region of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2019-05-27; First posted 2019-06-04 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Social Anxiety
Keywords: Social Anxiety Disorder; Virtual Reality; Exposure Therapy; Randomized Controlled Trial
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy; Implosive Therapy; Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: An equal number of participants will be assigned to each group, but at the end of treatment participants in the third group will be randomly re-allocated to one of the two former groups
Masking Description: Assignment will be kept blind for participants and clinicians until the first exposure session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Exposure Therapy (Experimental): VRET will include 360° videos with three scenarios a) riding a bus, b) going to a school cafeteria and c) a job interview. These scenarios were chosen based on clinical experience and frequently reported difficult situations in the literature . The order of the scenarios is jointly decided by the patient and therapist. In the videos the patients can make choices which determine the further course of the exposure scenario. For example, in the bus scenario the information system is out of order. Therefore, the patient has to ask the driver to announce, when they are at a particular stop. Depending on whether or not the patient decides to do so, the video will skip to one of two alternative continuations of the scenario. During the exposures the therapist will also motivate the patient towards acting in ways they consider unacceptable to provoke fear of ridicule, and make the patient act against him or her excessively rigid rules for social interaction to observe the consequences.
  Interventions: Behavioral: Cognitive Behavioral Therapy with Exposure therapy
- In Vivo Exposure Therapy (Active Comparator): In vivo exposure consists of role-playing and guided exposure either inside or outside the therapist's office with active modelling from the therapist in early sessions. Staff members are called upon to conduct exposure. Similarly to the VRET during in vivo exposure the therapist will motivate the patient towards acting in ways they consider unacceptable.
  Interventions: Behavioral: Cognitive Behavioral Therapy with Exposure therapy
- Virtual Reality Relaxation Therapy (Placebo Comparator): VR relaxation therapy will consist of a VR scenario of swimming with dolphins, created by the dolphin swim club (www.thedolphinswimclub.com). Swimming with real wild dolphins has been shown to have a positive effect on anxiety, although not specifically on SAD
  Interventions: Behavioral: Relaxation Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy with Exposure therapy — Treatment will be conducted for 10 consecutive weekly 60 min sessions. In the first two treatment conditions sessions are scheduled as follows: Session one: Building a therapeutic alliance and psycho-education about social anxiety and safety and avoidance behaviors. Session two to four: Cognitive restructuring. Session five to nine: Exposure in either in vivo or VR. Session 10: Relapse prevention. Sessions one to four and ten are identical in the two of three treatment arms.
  Arms: In Vivo Exposure Therapy; Virtual Reality Exposure Therapy
Behavioral: Relaxation Therapy — Relaxation Therapy
  Arms: Virtual Reality Relaxation Therapy

SUMMARY:
Social Anxiety Disorder (SAD) is classified as a phobic (anxious) disorder in which the patient experiences anxiety in social interactions, during which he or she might be judged or socially evaluated by others. SAD has an estimated lifetime prevalence of 3-13%, but remains under-treated. The recommended psychological treatment for SAD is is the exposure technique imbedded in Cognitive Behavioral Therapy (CBT). Traditionally exposure has taken place either in vivo or through imaginary exposure. In vivo has shown to be most effective, but it is costly and time-consuming and situational elements, such as the reaction of others, are difficult to control. Recently, researchers and clinicians have started to use Virtual Reality (VR) to overcome such difficulties. Compared to traditional methods VR-based Exposure has several advantages mainly based on increased control.

Meta-analyzes have found superior effect of CBT with VR-based Exposure compared to imaginary exposure, and similar effects when compared to in vivo exposure, with a recent study finding superior effect of VR-based Exposure compared to in vivo. The current evidence thus supports the clinical efficacy of CBT with VR-based Exposure. However, the meta-analyzes include a total of only six randomized controlled trials (RCTs) and only four of these compare CBT with VR-based Exposure to both an in vivo and a control group.

The aims of the current study are to develop a complete program of CBT with VR exposure based on 360° videos for adults suffering from SAD, and to evaluate the treatment effect on SAD symptoms.

The study is designed as a three arm RCT comparing 1) a group receiving CBT with VR-based Exposure, 2) a group receiving CBT with in vivo exposure and 3) a group receiving VR relaxation.

CBT with VR-based Exposure, will include 360° videos with three different scenarios In Vivo Exposure Therapy consists of role-playing and guided exposure either inside or outside the therapist's office.

VR Relaxation Therapy consists of a VR scenario of swimming with dolphins. Treatment will last 10 weeks and there will be a 6 months follow-up.

. It is hypothesized that

* CBT with VR-based Exposure will reduce symptoms of SAD
* CBT with VR-based Exposure will be more effective than both CBT with in vivo exposure and VR relaxation therapy at the end of treatment
* An effect on symptom reduction will sustain at the 6 months follow-up

DETAILED DESCRIPTION:
Introduction Social Anxiety Disorder (SAD) is a common yet underreported mental disorder with an estimated lifetime prevalence of 3-13%, and low rates of spontaneous remission. Patients with SAD experience intense and persistent fear in social interactions, during which he or she might be judged or negatively evaluated by others (e.g. public speaking, shopping). Symptoms include overwhelming bodily symptoms, such as sweating, trembling and increased heart rate, leading to avoidance of social situations (e.g. education, work) and significant functional impairment. SAD is highly debilitating, with the majority of socially anxious persons reporting numerous problems in individual and social adjustment, and with associated impairment in academic and professional functioning. Moreover, SAD often co-occurs with other psychiatric conditions such as mood disorders and substance use disorders, and is significantly associated with suicidal ideation. Despite its frequency and severity, only between one third and half of people with SAD seek treatment.

The recommended psychological treatment for SAD is the exposure technique imbedded in Cognitive Behavioral Therapy (CBT). CBT for SAD combines cognitive restructuring with exposure. In exposure-based therapy, exposures to social situations are used to test the patient's predictions about the danger in a particular situation. Further, it helps the patient develop new, realistic mental representations associated with the feared stimuli. Patients with SAD often have excessively high standards for social performance, and a strong fear of ridicule. Thus, it can be particularly helpful to encourage patients to behave in ways that they would consider unacceptable. i.e. intentionally acts against their excessively rigid rules for social interaction while observing the consequences.

Exposure has traditionally taken place as either:

1. In vivo: directly facing the feared situation.
2. Imaginary exposure: imagining the feared situation (can be facilitated through pictures or videos).

In vivo exposure is effective, but is costly, time-consuming and situational elements, such as the reaction of others, are difficult to control. Furthermore, many patients are rather unwilling to expose themselves to the real situation since it is considered too frightening. Furthermore, there is a risk of encountering familiar people revealing that the person is in therapy. Conversely, imaginary exposure may lack realism and intensity , and can be difficult for people who are unable to imagine vividly, avoid imagining their phobia-inducing situations, or tend to overwhelm themselves with images. Recently, researchers and clinicians have started to use Virtual Reality (VR) to overcome these difficulties.

Virtual reality based exposure

VR immerse the user in a computer generated or video-based virtual environment, using computer graphics or 360° videos. Studies on the effect of VR-based treatment for different types of phobias (e.g. agoraphobia and fear of flying) have revealed great potential, and a recent study showed that 76% of participants preferred VR-based exposure over in vivo exposure. Compared to traditional exposure methods VR-based exposure does have several advantages:

Virtual exposure scenarios can be very similar to real life situations, and it is possible to control and regulate situational factors, such as difficulty for the patient and the reactions of other people in the VE.

Exposure scenarios can be presented to the patients, while still in the comfort and safety of a therapeutic room, and exposure can be stopped at any time in case of excessive emotional activation.

VR-sessions often requires less time than in vivo sessions, and can be planned more flexibly and for less costs

Seven meta-analyzes have been published on CBT with VR-based exposure for anxiety, and six of these include studies on SAD. All found superior effect of CBT with VR-based exposure compared to imaginary exposure, and similar effects when compared to in vivo exposure, with a recent study finding superior effect of CBT with VR-based exposure even when compared to in vivo. Treatment effects have been shown to persist over a number of years, and a recent meta-analysis found persistence of benefits of treatment after CBT with VR-based exposure to be as good as face-to-face therapy. Furthermore, a meta-analysis found that the benefits carry over to real life, and that CBT with VR-based exposure leads to significant behavior change in real-life situations, even if this did not include SAD specific studies. The current evidence thus supports the clinical efficacy of CBT with VR-based exposure, and it is suggested that if the potential of VR is fully explored it might be more effective than in vivo.

Aims and hypotheses

The aims of the current study are to develop a complete program of CBT with VR exposure based on 360° videos for adult patients suffering from SAD, and to evaluate the treatment effect on SAD symptoms. We plan to compare a group receiving CBT with VR-based exposure immersed in an environment based on 360 videos stimuli to a group receiving CBT with in vivo exposure and a group receiving VR relaxation treatment. Having VR relaxation treatment as control group is methodologically superior to a comparison to a waiting list and controls for any placebo effect.

It is hypothesized that:

CBT with VR-based exposure will significantly reduce symptoms of SAD CBT with VR-based exposure will be more effective than both CBT with in vivo exposure and VR relaxation therapy at the end of treatment An effect on symptom reduction will sustain at 6 months follow-up

METHOD Design The study is designed as a three arm randomized controlled trial comparing a group receiving CBT with VR-based exposure, a group receiving CBT with in vivo exposure and a group receiving VR relaxation.

Participants and recruitment

Patients are recruited from the mental health services in the Region of Southern Denmark and from the Internet clinic at the Centre for Telepsychiatry (CTP). Patients are also recruited from the municipalities in this Danish region. Case managers at the job centers in the municipalities will be trained by the research leader to identify potential patients. Furthermore, we will advertise on the homepages for the CTP, for the Region of Southern Denmark, and at a national health website sundhed.dk

Participants will receive written information material and be asked to complete an online version of the Social Interaction Anxiety Scale (SIAS). If SAD score is above cut-off they are invited to a meeting conducted either at the CTP or through video call for oral information and diagnostic assessment. All potential participants will have their diagnoses discussed at weekly clinical conference. Those who meet the inclusion criteria will be offered participation and be asked to sign an informed consent statement.

Study data will be collected and managed using the Research Electronic Data Capture (REDCap) tools hosted at the mental health services in the Region of Southern Denmark. REDCap is a secure, state-of-the-art web-based application designed to support data capture for research studies.

Randomization and blinding Patients are randomly assigned (by gender, age and baseline severity of SAD) to one of the following three arms in ratio 1:1:1 via the computerized randomization function in REDCap: 1) Individual CBT with VR-based exposure in session 2) Individual CBT with in vivo exposure in session or 3) Individual VR relaxation therapy. Assignment will be kept blind for patients and clinicians until the first exposure session. An equal number of patients will be assigned to each group, but at the end of treatment patients in the third group will be randomly re-allocated to one of the two former groups. This reallocation is done to reduce the total number of patients needed to be recruited, and to avoid the ethical problem of not offering effective treatment. Six months after end of treatment the patients in group 1 and 2 will be re-assessed. There will not be a follow-up assessment of the patients in group 3, as they are re-allocated after week 10.

Intervention Treatment will be conducted by two clinical psychologists who will receive supervision every second week. Ten percent of the sessions will be audio recorded to ensure adherence to the treatment manual.

Assessment Diagnostic assessment will be conducted with the short version of the Present State Examination (PSE) supplemented with the anxiety section from the full version. PSE is a semi-structured interview, intended to provide an objective evaluation of present mental disorders. It contains 140 items, each scored on a 3-point or 4-point scale.

Primary and secondary outcome measures The primary outcome is severity of SAD, with the Social Interaction Anxiety Scale (SIAS). The scale has been used and validated in international research, has good psychometric properties , and focus on the interactional aspects of SAD, more so than on situations in which the person may be observed or scrutinized by others.

As a measure of general functioning we use the EQ-5D-5L. To study the practical and financial resources needed for exposure sessions, we include the questionnaire 'Specific Work for Exposure Applied in Therapy' (SWEAT). The Working Alliance Inventory-Short Revised (WAI-SR) is a measure of the therapeutic alliance .

Other measures Symptoms of ADHD and severity of autism spectrum disorder (ASD) characteristics will be assessed at baseline with the adult ADHD self-report scale (ASRS v1.1) and social responsiveness scale (SRS-2) respectively . Alcohol and drug use will be assessed with the Alcohol Use Disorders Identification Test (AUDIT) and the drug use disorders identification test (DUDIT) respectively. Depressive symptoms will be assessed with the Beck Depression Inventory-II (BDI-II) , which is the most widely used instrument for detecting depression.

Consent to participate All participants receive both written and oral information about the project and signed written informed consent is provided by all participants in the study.

Modification of the Protocol Any modifications to the protocol which may impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, patient population, sample sizes, study procedures, or significant administrative aspects will require a formal amendment to the protocol. Such amendment will be agreed upon by the authors of the current protocol, and approved by the Ethics Committee. Administrative changes of the protocol are minor corrections and/or clarifications that have no effect on the way the study is to be conducted. These administrative changes will be agreed upon by the authors of the current protocol, and will be documented in a memorandum.

Dissemination of results The primary results will be published in a relevant scientific journal independent of outcome. CONSORT guidelines will be respected, and both negative and positive results will be published.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend the Danish language
* ≥18 years
* Fulfill the diagnostic criteria for SAD according to ICD-10 (F40.1) or ICD-11 (6B04)

Exclusion Criteria:

* Previously diagnosed with psychosis, Autism Spectrum Disorder or severe depression.
* Participating in other psychotherapeutic treatments during the study
* Substance dependence disorder
* Severe cyber-sickness (corresponding to driving sickness).
* If on medication, medication must be stable for 6 months prior to the study and during the study (i.e., no change).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
change in Social Interaction Anxiety Scale (SIAS) | change from baseline to week 10
  Severity of Social Anxiety Disorder. SIAS is a measure of anxiety in social interactional situations and consist of 20 items scored 0-4. The total score range from 0-80 with a score higher than 43 indicating that SAD is probable

SECONDARY OUTCOMES:
Specific Work for Exposure Applied in Therapy (SWEAT). | week 10
  The practical and financial resources needed for exposure sessions. SWEAT measures cost and efforts required to conduct exposure sessions. The questionnaire consists of 11 items
change in EQ-5D-5L | change from baseline to week 10
  General functioning. EQ-5D-5L is a standardized instrument for measuring generic health status.
The Working Alliance Inventory-Short Revised (WAI-SR) | week 10
  The therapeutic alliance. WAI-SR assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond.

CONTACTS AND LOCATIONS:
Overall Officials: Per Trads Ørskov, PhD, Principal Investigator — Region of Southern Denmark
Locations (1):
- Centre for Telepsychiatry, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso J, Lepine JP; ESEMeD/MHEDEA 2000 Scientific Committee. Overview of key data from the European Study of the Epidemiology of Mental Disorders (ESEMeD). J Clin Psychiatry. 2007;68 Suppl 2:3-9. PMID 17288501
- [Background] Craske MG, Stein MB. Anxiety. Lancet. 2016 Dec 17;388(10063):3048-3059. doi: 10.1016/S0140-6736(16)30381-6. Epub 2016 Jun 24. PMID 27349358
- [Background] Stein DJ, Lim CCW, Roest AM, de Jonge P, Aguilar-Gaxiola S, Al-Hamzawi A, Alonso J, Benjet C, Bromet EJ, Bruffaerts R, de Girolamo G, Florescu S, Gureje O, Haro JM, Harris MG, He Y, Hinkov H, Horiguchi I, Hu C, Karam A, Karam EG, Lee S, Lepine JP, Navarro-Mateu F, Pennell BE, Piazza M, Posada-Villa J, Ten Have M, Torres Y, Viana MC, Wojtyniak B, Xavier M, Kessler RC, Scott KM; WHO World Mental Health Survey Collaborators. The cross-national epidemiology of social anxiety disorder: Data from the World Mental Health Survey Initiative. BMC Med. 2017 Jul 31;15(1):143. doi: 10.1186/s12916-017-0889-2. PMID 28756776
- [Background] Stein MB, Stein DJ. Social anxiety disorder. Lancet. 2008 Mar 29;371(9618):1115-25. doi: 10.1016/S0140-6736(08)60488-2. PMID 18374843
- [Background] Kampmann IL, Emmelkamp PM, Morina N. Meta-analysis of technology-assisted interventions for social anxiety disorder. J Anxiety Disord. 2016 Aug;42:71-84. doi: 10.1016/j.janxdis.2016.06.007. Epub 2016 Jun 18. PMID 27376634
- [Background] Bouchard S, Dumoulin S, Robillard G, Guitard T, Klinger E, Forget H, Loranger C, Roucaut FX. Virtual reality compared with in vivo exposure in the treatment of social anxiety disorder: a three-arm randomised controlled trial. Br J Psychiatry. 2017 Apr;210(4):276-283. doi: 10.1192/bjp.bp.116.184234. Epub 2016 Dec 15. PMID 27979818
- [Derived] Clemmensen L, Bouchard S, Rasmussen J, Holmberg TT, Nielsen JH, Jepsen JRM, Lichtenstein MB. STUDY PROTOCOL: EXPOSURE IN VIRTUAL REALITY FOR SOCIAL ANXIETY DISORDER - a randomized controlled superiority trial comparing cognitive behavioral therapy with virtual reality based exposure to cognitive behavioral therapy with in vivo exposure. BMC Psychiatry. 2020 Jan 30;20(1):32. doi: 10.1186/s12888-020-2453-4. PMID 32000725